CLINICAL TRIAL: NCT00867646
Title: Comparison Study of CoaguChek XS Prothrombin Time and Laboratory Innovin PT by NTUH Lab Medicine
Brief Title: Comparison Study of CoaguChek XS PT and Laboratory Innovin PT by NTUH Lab Medicine
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Chiang, Fu-Tien/ Director of Laboratory Medicine, National Taiwan University Hospital
Other Study IDs: 20080418R
Record Dates: First submitted 2008-08-01; First posted 2009-03-24 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2009-12

CONDITIONS: Deep Vein Thrombosis
Keywords: PT; DVT
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Comparison Study of CoaguChek XS PT and Laboratory Innovin PT by NTUH Lab Medicine

DETAILED DESCRIPTION:
This trial is going to proceed in two phases: Familiarization Phase and Evaluation Phase. The Preliminary Comparison Study consists of ten (10) patients being tested with the CoaguChek system and the laboratory reference method. This preliminary study is intended to help familiarize the operator with the dosing of the CoaguChek XS PT strips and to serve as an indicator as to whether some of the variables. Evaluation Phase consists of testing seventy (70) patient samples with the CoaguChek XS system and with the laboratory method.

ELIGIBILITY:
Inclusion Criteria:

* Warfarin continuously treated patients

Exclusion Criteria:

* Warfarin recently discontinuous treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 70 Warfarin teated patients
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2008-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Comparison of the PTINR measured by Coaguchek and laboratory CA1500 | 2 Months

CONTACTS AND LOCATIONS:
Overall Officials: Chiang Fu-Tien, PhD, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan